CLINICAL TRIAL: NCT00327470
Title: A 102-Week, Open Label, Multicenter Trial To Investigate The Efficacy Of Macugen For The Preservation Of Visual Function In Subjects With Neovascular Age-Related Macular Degeneration (AMD) And To Assess The Benefit Of Treating Early Choroidal Neovascularization (CNV).
Brief Title: An Open Label Trial to Investigate Macugen for the Preservation of Visual Function in Subjects With Neovascular AMD
Acronym: PERSPECTIVES
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A5751017
Record Dates: First submitted 2006-05-17; First posted 2006-05-18 (Estimated); Results first posted 2010-12-17 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2011-01

CONDITIONS: Age Related Macular Degeneration (AMD); Macular Degeneration; Choroidal Neovascularization (CNV)
Keywords: neovascular age related macular degeneration; choroidal neovascularization
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — pegaptanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open Label (Experimental)
  Interventions: Drug: Pegaptanib Sodium 0.3 mg

INTERVENTIONS:
Drug: Pegaptanib Sodium 0.3 mg — Pegaptanib Sodium dosed every 6 weeks in affected eye.

SUMMARY:
The purpose of this study is to determine the benefits of treating subjects with neovascular age-related macular degeneration (AMD) at an earlier stage of choroidal neovascularization (CNV) as compared to those with established CNV. Additionally, the study would like to determine the efficacy of Macugen in preserving visual function in those subjects having CNV secondary to neovascular AMD.

DETAILED DESCRIPTION:
A decision was made by the sponsor (08 May 2009) to terminate this study early; the study had achieved the primary objective prior to termination. This study was not terminated due to safety reasons.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of neovascular AMD in at least one eye. In subjects with bilateral neovascular AMD, only one eye would be eligible for enrollment
* Baseline visual acuity of greater than or equal to 20/320, or better than 25 ETDRS letters in the study eye

Exclusion Criteria:

* Previous treatment for CNV secondary to AMD, including any prior PDT with verteporfin, thermal laser photocoagulation, external beam radiation or transpupillary thermotherapy to the study eye
* Subjects having subfoveal fibrosis/ scar or atrophy representing > 25% of the total lesion size

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2006-07; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (48):
- Austria (3):
  - Pfizer Investigational Site, Graz
  - Pfizer Investigational Site, Innsbruck
  - Pfizer Investigational Site, Vienna
- Belgium (2):
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Liège
- Canada (5):
  - Pfizer Investigational Site, Victoria, British Columbia
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
- Czechia (2):
  - Pfizer Investigational Site, Olomouc
  - Pfizer Investigational Site, Prague
- Pfizer Investigational Site, Glostrup Municipality, Denmark
- Pfizer Investigational Site, Kuopio, Finlad, Finland
- France (6):
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Nancy
  - Pfizer Investigational Site, Nantes
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Saint-Etienne
  - Pfizer Investigational Site, Tours
- Germany (4):
  - Pfizer Investigational Site, Dortmund
  - Pfizer Investigational Site, Freiburg im Breisgau
  - Pfizer Investigational Site, Halle
  - Pfizer Investigational Site, Münster
- Pfizer Investigational Site, Athens, Greece
- Italy (4):
  - Pfizer Investigational Site, Ancona
  - Pfizer Investigational Site, Bari
  - Pfizer Investigational Site, Florence
  - Pfizer Investigational Site, Milan
- Poland (4):
  - Pfizer Investigational Site, Gdansk
  - Pfizer Investigational Site, Katowice
  - Pfizer Investigational Site, Poznan
  - Pfizer Investigational Site, Warsaw
- Portugal (3):
  - Pfizer Investigational Site, Coimbra
  - Pfizer Investigational Site, Lisbon
  - Pfizer Investigational Site, Porto
- Spain (4):
  - Pfizer Investigational Site, Alicante, Alicante
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Santiago de Compostela, La Coruña
  - Pfizer Investigational Site, Valencia, Valencia
- Turkey (Türkiye) (2):
  - Pfizer Investigational Site, Ankara
  - Pfizer Investigational Site, Istanbul
- United Kingdom (6):
  - Pfizer Investigational Site, Edinburgh, Midlothian
  - Pfizer Investigational Site, Aberdeen, Scotland
  - Pfizer Investigational Site, Belfast
  - Pfizer Investigational Site, Bristol
  - Pfizer Investigational Site, Leeds
  - Pfizer Investigational Site, Southampton

REFERENCES:
- [Derived] Chakravarthy U, Staurenghi G, Kwok K, Tressler CS, Buggage R; PERSPECTIVES Study Group. Treating early choroidal neovascularisation with pegaptanib sodium in patients with neovascular age-related macular degeneration: findings of the PERSPECTIVES study. Br J Ophthalmol. 2012 Oct;96(10):1351-4. doi: 10.1136/bjophthalmol-2011-301444. Epub 2012 Aug 7. No abstract available. PMID 22872673
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5751017&StudyName=An%20Open%20Label%20Trial%20to%20Investigate%20Macugen%20for%20the%20Preservation%20of%20Visual%20Function%20in%20subjects%20with%20Neovascular%20AMD

RESULTS

PARTICIPANT FLOW:
Groups:
- Early Age-related Macular Degeneration (AMD): Subjects with early choroidal neovascularization (CNV) lesions were distinguished from subjects with established CNV lesions based on the stage of evolution of their CNV as determined by fluorescein angiography and, where available, indocyanine green angiography as assessed by the investigator at Baseline. Subjects with early CNV lesions were treated in the study eye with Macugen (0.3 milligram [mg]) every 6 weeks for 48 weeks. All subjects completing the first year of therapy (54 weeks [ie, 6 weeks after treatment at Week 48]) continued treatment in the second year of the study (Weeks 54 to 102), with Macugen (0.3 mg) administered every 12 weeks (ie, Weeks 60, 72, 84, and 96).
- Established AMD: Subjects with established CNV lesions (as assessed by the investigator at Baseline) were treated in the study eye with Macugen (0.3 mg) every 6 weeks for 48 weeks. All subjects completing the first year of therapy (54 weeks [ie, 6 weeks after treatment at Week 48]) continued treatment in the second year of the study (Weeks 54 to 102), with Macugen (0.3 mg) administered every 12 weeks (ie, Weeks 60, 72, 84, and 96).
Period: Overall Study
Arm/Group | Early Age-related Macular Degeneration (AMD) | Established AMD
Started | 107 | 181
Treated | 107 | 179
Completed | 78 | 118
Not Completed | 29 | 63
Not completed — Randomized, but not treated | 0 | 2
Not completed — Adverse Event | 9 | 14
Not completed — Lack of Efficacy | 7 | 19
Not completed — Other | 5 | 9
Not completed — Lost to Follow-up | 1 | 3
Not completed — Withdrawal by Subject | 6 | 12
Not completed — Death | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Early AMD: Subjects with early CNV lesions (assessed by the investigator at Baseline) were treated in the study eye with Macugen (0.3 mg) every 6 weeks for 48 weeks. All subjects completing the first year of therapy (54 weeks [ie, 6 weeks after treatment at Week 48]) continued treatment in the second year of the study (Weeks 54 to 102), with Macugen (0.3 mg) administered every 12 weeks (ie, Weeks 60, 72, 84, and 96).
- Total: Total of all reporting groups
Arm/Group | Early AMD | Established AMD | Total
Number analyzed (Participants) | 107 | 179 | 286
Age, Customized [Number; unit: Participants]
  45 through 64 years | 12 | 24 | 36
  >= 65 years | 95 | 155 | 250
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 108 | 167
  Male | 48 | 71 | 119

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline Through Week 54 in Distance Visual Acuity (VA) in Subjects With Early and Established CNV Lesions
Description: The investigator assessed the best-corrected VA obtained by a protocol refraction using the retroilluminated modified Ferris-Bailey Early Treatment of Diabetic Retinopathy Study (ETDRS) charts recorded at a 2-meter distance from the chart. Distance VA was expressed as an ETDRS score (number of letters correctly read): the proportion of subjects losing >=30 letters or <15 letters from Baseline, gaining >=0 or >=15 letters from Baseline. The mean change in VA from Baseline at Week 54 was assessed.
Time Frame: Baseline through Week 54
Population: The modified intent-to-treat (MITT) population included all subjects in the safety population who had a Baseline distance VA measurement and at least 1 post-Baseline VA measurement. Last observation carried forward (LOCF). Note: the number of participants analyzed refers to the number of subjects who had data that could be analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Early AMD | Established AMD
Number analyzed (Participants) | 107 | 178
Scores on a scale | -4.30 (14.57) | -5.51 (15.08)

2. Secondary Outcome: Mean Change From Baseline in Distance VA in Subjects With Early and Established CNV Lesions
Description: The investigator assessed the best-corrected VA obtained by a protocol refraction using the retroilluminated modified Ferris-Bailey ETDRS charts recorded at a 2-meter distance from the chart. Distance VA was expressed as an ETDRS score (number of letters correctly read): the proportion of subjects losing >=30 letters or <15 letters, gaining >=0 or >=15 letters. The mean changes in VA from Baseline/Week 102 and Week 52/102 were assessed.
Time Frame: Baseline through Week 102, Week 54 through Week 102
Population: MITT LOCF; Note: the number of participants analyzed refers to the number of subjects who had data that could be analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Early AMD | Established AMD
Number analyzed (Participants) | 107 | 178
Scores on a scale
  Baseline through Week 102 | -7.91 (16.14) | -8.95 (17.34)
  Week 54 through Week 102 | -3.61 (9.83) | -3.44 (9.81)

3. Secondary Outcome: Mean Change From Baseline in Near VA in Subjects With Early and Established CNV Lesions
Description: Near VA was measured with the modified Bailey-Lovie near-word reading charts at a distance of 25 centimeters using a +3.50 reading addition worn over the protocol refraction providing the best-corrected distance VA. The reading charts test the smallest word size identifiable from 0.0 logarithmic of the minimum angle of resolution (logMAR) to 1.6 logMAR. logMAR is the logarithm of the minimum angle of resolution. The ideal is 0.0 and represents 20/20 Snellen acuity. logMAR values >0.00 indicate vision poorer than ideal and values <0.0 indicate vision greater than ideal.
Time Frame: Baseline through Week 54, Baseline through Week 102
Population: MITT LOCF. Note: the number of participants analyzed refers to the number of subjects who had data that could be analyzed. n=number of subjects with evaluable data.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Early AMD | Established AMD
Number analyzed (Participants) | 107 | 178
Scores on a scale
  Baseline through Week 54 (n=104, n=172) | 0.10 (0.27) | 0.15 (0.32)
  Baseline through Week 102 (n=105, n=172) | 0.19 (0.34) | 0.22 (0.36)

4. Secondary Outcome: Mean Change in Reading Speed
Description: For assessment of reading speed, subjects were asked to read a print steadily, without stopping or interruption, at a comfortable pace. On commencing reading, a timer was activated. The timer was stopped when the subject had finished reading all of the words on the chart or at 2 minutes, whichever was sooner. Only the total number of words read correctly was recorded. The time recorded for the reading speed test was the time required for the subject to finish reading all of the words on the chart in minutes and seconds (maximum 2 minutes).
Time Frame: Baseline through Week 54, Baseline through Week 102, and Week 54 through Week 102
Population: MITT LOCF; Note: the number of participants analyzed refers to the number of subjects who had data that could be analyzed. n=number of subjects with evaluable data.
Measure: Mean (Standard Deviation); unit: Correctly read words per minute
Arm/Group | Early AMD | Established AMD
Number analyzed (Participants) | 107 | 178
Correctly read words per minute
  Baseline through Week 54 (n=92, n=151) | -9.15 (28.78) | -10.98 (22.31)
  Baseline through Week 102 (n=94, n=152) | -17.81 (28.48) | -12.23 (32.08)
  Week 54 through Week 102 (n=93, n=152) | -8.43 (18.06) | -1.15 (23.77)

5. Secondary Outcome: Mean Change From Baseline in Contrast Sensitivity
Description: Contrast sensitivity was measured using the Pelli-Robson chart at 1 meter. Subjects were tested for contrast sensitivity using +0.50 addition over the protocol refraction providing the best-corrected distance VA. Contrast sensitivity was recorded as the log of the faintest triplet for which 2 of the 3 letters were read correctly.
Time Frame: Baseline through Week 54, Baseline through Week 102
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Correctly read letters
Arm/Group | Early AMD | Established AMD
Number analyzed (Participants) | 107 | 178
Correctly read letters
  Baseline through Week 54 (n=93, n=152) | -0.06 (0.26) | -0.03 (0.33)
  Baseline through Week 102 (n=94, n=152) | -0.16 (0.37) | -0.09 (0.39)

6. Secondary Outcome: Mean Change in National Eye Institute - Visual Functioning Questionnaire (NEI-VFQ-25) Composite Score
Description: Subject reported vision-related functioning and Quality of Life (QoL) as measured using the 25 item NEI-VFQ-25. Items are grouped as the following - Composite: mean score items 1-25; General Health: item 1; General Vision: item 2; Ocular Pain: 4,19; Near Vision: 5,6,7; Distance Vision: 8,9,14; Social Functioning: 11,13; Mental Health Activities: 3,21,22,25; Role Difficulties: 17,18; Dependency: 20,23,24; Driving: 15c,16, 16a; Color Vision: 12; Peripheral Vision: 10. A positive change represents an increase in function/health, a negative change represents a decrease in function/health.
Time Frame: Baseline through Week 54, Baseline through Week 102, and Week 54 through Week 102
Population: MITT. Note: the number of participants analyzed refers to the number of subjects who had data that could be analyzed. n=number of subjects with evaluable data.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Early AMD | Established AMD
Number analyzed (Participants) | 107 | 178
Scores on a scale
  Baseline through Week 54 (n=90, n=146) | -1.54 (12.946) | -1.03 (13.264)
  Baseline through Week 102 (n=67, n=111) | -4.57 (14.410) | -1.65 (12.569)
  Week 54 through Week 102 (n=64, n=115) | -2.74 (9.655) | -2.48 (9.473)

7. Secondary Outcome: Mean Change in Euro QoL Questionnaire (EQ-5D) Score
Description: The EQ-5D is a validated, standardized QoL instrument assessing general health status based on the preference of a UK general population. It consists of two sections: a 100-point visual analog scale (VAS) and a descriptive system that contains five attributes (mobility, self-care, usual activities, pain or discomfort, and anxiety or depression) with three levels per attribute ("no problem", "some problems" and "extreme problems"). A subject's responses to these domains were mapped to a corresponding score of the EQ-5D index.
Time Frame: Baseline through Week 54, Baseline through Week 102, and Week 54 through Week 102
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Early AMD | Established AMD
Number analyzed (Participants) | 107 | 178
Scores on a scale
  Baseline through Week 54 (n=90, n=146) | -0.00 (0.260) | -0.01 (0.227)
  Baseline through Week 102 (n=67, n=111) | -0.04 (0.267) | -0.04 (0.207)
  Week 54 through Week 102 (n=64, n=115) | -0.01 (0.271) | -0.03 (0.213)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Early AMD | Established AMD
Serious Adverse Events (participants affected / at risk) | 23/107 | 32/179
Other Adverse Events (participants affected / at risk) | 68/107 | 120/179
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Early AMD (N=107) | Established AMD (N=179)
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 3 | 0
Angina unstable (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 2
Bradycardia (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 1
Eye haemorrhage (Eye disorders) | 0 | 2
Iridocyclitis (Eye disorders) | 0 | 1
Open angle glaucoma (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1
Uveitis (Eye disorders) | 0 | 2
Visual acuity reduced (Eye disorders) | 0 | 1
Vitritis (Eye disorders) | 0 | 1
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Injection site injury (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Endophthalmitis (Infections and infestations) | 2 | 2
Gastroenteritis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 3
Loss of consciousness (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Eye operation (Surgical and medical procedures) | 1 | 0
Meniscus operation (Surgical and medical procedures) | 0 | 1
Arterial thrombosis limb (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early AMD (N=107) | Established AMD (N=179)
Anaemia (Blood and lymphatic system disorders) | 0 | 4
Splenic lesion (Blood and lymphatic system disorders) | 1 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 2
Cardiac failure (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1
Corneal dystrophy (Congenital, familial and genetic disorders) | 1 | 0
Deafness (Ear and labyrinth disorders) | 0 | 2
Vertigo (Ear and labyrinth disorders) | 3 | 2
Anterior chamber cell (Eye disorders) | 3 | 3
Anterior chamber flare (Eye disorders) | 1 | 0
Anterior chamber pigmentation (Eye disorders) | 2 | 0
Aphakia (Eye disorders) | 1 | 0
Blepharitis (Eye disorders) | 2 | 2
Blepharitis allergic (Eye disorders) | 0 | 1
Blindness (Eye disorders) | 2 | 2
Blindness transient (Eye disorders) | 0 | 1
Blindness unilateral (Eye disorders) | 3 | 0
Cataract (Eye disorders) | 2 | 4
Cataract nuclear (Eye disorders) | 1 | 1
Cataract subcapsular (Eye disorders) | 0 | 1
Chalazion (Eye disorders) | 1 | 2
Choroidal neovascularisation (Eye disorders) | 1 | 6
Ciliary body haemorrhage (Eye disorders) | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 17 | 16
Conjunctival hyperaemia (Eye disorders) | 7 | 4
Conjunctival oedema (Eye disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 7 | 8
Corneal deposits (Eye disorders) | 0 | 1
Corneal disorder (Eye disorders) | 2 | 2
Corneal epithelium defect (Eye disorders) | 10 | 4
Corneal erosion (Eye disorders) | 0 | 3
Corneal oedema (Eye disorders) | 5 | 7
Corneal opacity (Eye disorders) | 0 | 2
Detachment of retinal pigment epithelium (Eye disorders) | 1 | 1
Dry eye (Eye disorders) | 1 | 3
Episcleritis (Eye disorders) | 1 | 0
Erythema of eyelid (Eye disorders) | 1 | 0
Eye discharge (Eye disorders) | 1 | 4
Eye disorder (Eye disorders) | 1 | 2
Eye haemorrhage (Eye disorders) | 3 | 2
Eye irritation (Eye disorders) | 1 | 5
Eye pain (Eye disorders) | 9 | 9
Eye pruritus (Eye disorders) | 1 | 0
Eyelid oedema (Eye disorders) | 1 | 1
Foreign body sensation in eyes (Eye disorders) | 4 | 0
Glaucoma (Eye disorders) | 1 | 1
Hyalosis asteroid (Eye disorders) | 0 | 1
Hyphaema (Eye disorders) | 0 | 1
Iridocyclitis (Eye disorders) | 0 | 3
Keratoconjunctivitis sicca (Eye disorders) | 0 | 1
Lacrimation increased (Eye disorders) | 6 | 2
Lens disorder (Eye disorders) | 1 | 0
Macular degeneration (Eye disorders) | 2 | 5
Maculopathy (Eye disorders) | 0 | 1
Metamorphopsia (Eye disorders) | 3 | 1
Myodesopsia (Eye disorders) | 6 | 4
Ocular hyperaemia (Eye disorders) | 3 | 3
Ocular hypertension (Eye disorders) | 0 | 2
Photophobia (Eye disorders) | 2 | 1
Photopsia (Eye disorders) | 1 | 1
Posterior capsule opacification (Eye disorders) | 1 | 3
Punctate keratitis (Eye disorders) | 0 | 2
Retinal artery spasm (Eye disorders) | 0 | 1
Retinal exudates (Eye disorders) | 1 | 1
Retinal haemorrhage (Eye disorders) | 3 | 9
Retinal oedema (Eye disorders) | 1 | 0
Retinal pigment epithelial tear (Eye disorders) | 1 | 1
Scleral haemorrhage (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 3 | 1
Visual acuity reduced (Eye disorders) | 2 | 9
Visual impairment (Eye disorders) | 2 | 4
Vitreous detachment (Eye disorders) | 3 | 1
Vitreous disorder (Eye disorders) | 7 | 6
Vitreous haemorrhage (Eye disorders) | 2 | 3
Vitreous opacities (Eye disorders) | 1 | 1
Vitritis (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Colitis (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 4
Dental caries (Gastrointestinal disorders) | 1 | 1
Dental plaque (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 2
Duodenogastric reflux (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 2
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Gingivitis (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1
Rectal prolapse (Gastrointestinal disorders) | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 0 | 2
Fatigue (General disorders) | 0 | 1
Influenza like illness (General disorders) | 1 | 0
Injection site haemorrhage (General disorders) | 1 | 4
Injection site irritation (General disorders) | 0 | 2
Injection site pain (General disorders) | 1 | 4
Injection site reaction (General disorders) | 2 | 0
Pain (General disorders) | 2 | 0
Polyp (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 0
Therapeutic response unexpected (General disorders) | 0 | 1
Hepatic cyst (Hepatobiliary disorders) | 1 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Liver disorder (Hepatobiliary disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 2
Hypersensitivity (Immune system disorders) | 0 | 1
Abscess (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 8
Candidiasis (Infections and infestations) | 0 | 1
Conjunctivitis bacterial (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 2
Dacryocystitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Eye infection (Infections and infestations) | 1 | 0
Fungal skin infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 2
Gastrointestinal fungal infection (Infections and infestations) | 1 | 0
Gingival infection (Infections and infestations) | 0 | 1
Herpes virus infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 1
Hordeolum (Infections and infestations) | 0 | 2
Incision site infection (Infections and infestations) | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 2 | 5
Keratitis herpetic (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 0 | 2
Lower respiratory tract infection (Infections and infestations) | 1 | 4
Nasopharyngitis (Infections and infestations) | 9 | 10
Otitis media (Infections and infestations) | 0 | 2
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Pulpitis dental (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 3
Tooth abscess (Infections and infestations) | 1 | 1
Tooth infection (Infections and infestations) | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 3 | 5
Urethritis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 3 | 1
Viral infection (Infections and infestations) | 1 | 0
Accidental exposure (Injury, poisoning and procedural complications) | 1 | 0
Cataract operation complication (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 2
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 3
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 2
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1
Ligament injury (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 1
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 2
Skeletal injury (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood glucose increased (Investigations) | 1 | 0
Blood pressure abnormal (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 0 | 3
Blood uric acid increased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1
Intraocular pressure decreased (Investigations) | 1 | 0
Intraocular pressure increased (Investigations) | 8 | 15
Ultrasound Doppler normal (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperhomocysteinaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Jaw cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 4
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 4
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Aphasia (Nervous system disorders) | 1 | 0
Balance disorder (Nervous system disorders) | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 4 | 7
Hemicephalalgia (Nervous system disorders) | 0 | 1
Hyperaesthesia (Nervous system disorders) | 2 | 0
Hypertonia (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Hyposmia (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0 (0)
Sciatica (Nervous system disorders) | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Trigeminal neuralgia (Nervous system disorders) | 0 | 1
Visual field defect (Nervous system disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 2
Confusional state (Psychiatric disorders) | 1 | 0
Depressed mood (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 2
Nervousness (Psychiatric disorders) | 0 | 1
Reading disorder (Psychiatric disorders) | 1 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal cyst (Renal and urinary disorders) | 0 | 1
Breast cyst (Reproductive system and breast disorders) | 1 | 0
Cystocele (Reproductive system and breast disorders) | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Abscess drainage (Surgical and medical procedures) | 0 | 1
Bladder neoplasm surgery (Surgical and medical procedures) | 1 | 0
Carpal tunnel decompression (Surgical and medical procedures) | 0 | 1
Curetting of chalazion (Surgical and medical procedures) | 0 | 1
Gingival operation (Surgical and medical procedures) | 1 | 0
Malignant tumour excision (Surgical and medical procedures) | 1 | 0
Tooth extraction (Surgical and medical procedures) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 0 | 3
Hypertension (Vascular disorders) | 5 | 10
Orthostatic hypotension (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0
Varicose vein (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.